CLINICAL TRIAL: NCT06614387
Title: Assessment of Safety and Efficacy of Vedolizumab in Pediatric Uclerative Colitis in Comparison With Standard Biological Therapy With Infliximab
Brief Title: Vedolizumab in Pediatric Ulcerative Colitis- Comparison With Infliximab
Acronym: VEDI-UC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JAROSLAW KIERKUS (Other)
Responsible Party: Sponsor-Investigator, JAROSLAW KIERKUS, Children's Memorial Health Institute, Children's Memorial Health Institute, Poland
Organization: Children's Memorial Health Institute, Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 2023-509775-16
Record Dates: First submitted 2024-09-17; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Vedolizumab; Infliximab; Children
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; vedolizumab

STUDY DESIGN:
Intervention Model Description: This is a multicenter, double-blind, randomized study to compare the safety, effectiveness and immunogenicity (antibodies against drug) of two biological drugs administered intravenously - vedolizumab (a drug not registered in pediatric patients) and infliximab (used as standard therapy), in pediatric patients with UC aged 6-18 years.
  Before enrollment to the study, informed consent must be obtained from the participant's legal guardian and, additionally, from the participant aged > 16 years before any procedures are performed.
Who Masked: Investigator
Masking Description: Allocation to therapeutic subgroups will be in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infliximab arm (Active Comparator): Patients meeting the inclusion criteria and not having any of the exclusion criteria will be randomized 1:1 to one of two study arms - intravenous administration of blinded active drug, infliximab or vedolizumab at weeks 0, 2, 6 and 14. Infliximab will be administered at a dose 5mg/kg body weight, and vedolizumab at a dose of 300 mg (body mass > 40 kg) and 10 mg/kg (body mass < 40kg).
  Interventions: Drug: Infliximab
- Vedolizumab arm (Experimental): Patients meeting the inclusion criteria and not having any of the exclusion criteria will be randomized 1:1 to one of two study arms - intravenous administration of blinded active drug, infliximab or vedolizumab at weeks 0, 2, 6 and 14. Infliximab will be administered at a dose 5mg/kg body weight, and vedolizumab at a dose of 300 mg (body mass > 40 kg) and 10 mg/kg (body mass < 40kg).
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Patients meeting the inclusion criteria and not having any of the exclusion criteria will be randomized 1:1 to one of two study arms - intravenous administration of blinded active drug, infliximab or vedolizumab at weeks 0, 2, 6 and 14. Infliximab will be administered at a dose 5mg/kg body weight, and vedolizumab at a dose of 300 mg (body mass > 40 kg) and 10 mg/kg (body mass < 40kg).
  Other Names: vedolizumab

SUMMARY:
This is a multicenter, double-blind, randomized study to compare the safety, effectiveness and immunogenicity (antibodies against drug) of two biological drugs administered intravenously - vedolizumab (a drug not registered in pediatric patients) and infliximab (used as standard therapy), in pediatric patients with UC aged 6-18 years.

Before enrollment to the study, informed consent must be obtained from the participant's legal guardian and, additionally, from the participant aged >16 years before any procedures are performed.

ELIGIBILITY:
Inclusion criteria

1. Participant aged 6 to 17 years at the time of study entry.
2. Patient with moderate or severe UC defined by the PUCAI score (min. 30 points) - diagnosed at least 1 month before the qualifying visit.
3. Individuals who failed to respond to, lost response to, or were intolerant to treatment with at least 1 of the following agents:

   * corticosteroids (prednisone at a dose of 1 mg/kg/day with a maximum dose of 40 mg/day, budesonide MMX 9 mg/day) or immunomodulating drugs (e.g. AZA, 6-MP, MTX).
   * in the case of 5 - ASA adrugs, corticosteroids, immunomodulating drugs, doses should remain stable for 2 weeks before administration of the study drug
4. Patients with UC proximal to the rectum (i.e. not limited to proctitis).
5. At least Mayo 1 on the endoscopic scale
6. People with up-to-date vaccinations in accordance with the preventive vaccination program adopted in Poland.

Exclusion criteria

1. People who have been previously treated with biological antiintegrin preparations, including: natalizumab, efalizumab, etrolizumab or addressin-1 adhesion molecule antagonists or rituximab.
2. People who were previously treated with vedolizumab.
3. People who were previously treated with infliximab
4. People with hypersensitivity or allergy to any of the excipients of vedolizumab or infliximab
5. People with active brain/meningeal disease, signs/symptoms or history of progressive multifocal leukoencephalopathy (PML) or any other serious neurological disorder including stroke, multiple sclerosis, brain tumor or neurodegenerative disease.
6. Individuals who currently require or are expected to require surgical intervention for UC during this study.
7. People who have had a partial or total colectomy or have a jejunostomy, ileostomy, colostomy, ileo-anal stoma, or known permanent intestinal stricture.
8. People with a current diagnosis of unspecified colitis.
9. People with clinical features suggestive of monogenic inflammatory bowel disease of very early onset.
10. The participant has other serious comorbidities that will limit his or her ability to complete the study.
11. Abnormal laboratory tests:

    * Hgb ≤ 8 g/dl
    * Leukocytes ≤ 2.5 x 10*9 cells/L
    * ALT and/or AST ≥ 3 x upper limit of normal
    * positive Quantiferon result
    * positive result in the stool sample for Clostridium difficile and/or stool culture for alarm pathogens Security

At every check-up visit:

* occurrence of: adverse events (AEs), serious AEs (serious AEs-SAEs), infections including opportunistic infections such as PML, liver damage, malignant tumors, infusion-related reactions and hypersensitivity
* vital signs, results of standard laboratory tests

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of biological treatment with vedolizumab and infliximab assessed/defined by the number of drug-related adverse events (AEs). | screening - Week 20
  Information on AEs will be collected on each check-up visit, physical examination, vital signs and lab test will be performed